CLINICAL TRIAL: NCT07054840
Title: Pain and Split-belt Motor Learning in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2334309
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Aging; Older Adults; Pain; Motor Learning
MeSH Terms: conditions — Pain | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Pain (No Intervention): Will receive no intervention.
- Pain (Experimental): Will receive capsaicin and heat combined to induce acute pain.
  Interventions: Behavioral: Capsaicin 0.1% cream combined with a heat pack and applied to the lower leg

INTERVENTIONS:
Behavioral: Capsaicin 0.1% cream combined with a heat pack and applied to the lower leg — Capsaicin is applied to the skin of one of the lower legs, then covered with a heat pack that is secured to the leg with self-adhesive wrap.
  Arms: Pain

SUMMARY:
The purpose of this research is to investigate the impact of acute pain, induced using an experimental pain paradigm of capsaicin paired with heat, on implicit locomotor learning and its retention in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-90 years old
* Self-identifying as generally medically healthy
* Able to read, write and speak English
* Able to provide informed consent and attend all testing sessions
* Willing to undergo the experimental pain paradigm, if selected

Exclusion Criteria:

* Resting heart rate < 50 or > 100 bpm
* Resting blood pressure < 90/60 or > 165/95
* Any history or current mental health condition, learning/developmental disability or cognitive impairment, including severe untreated ADD/ADHD, severe untreated anxiety, severe untreated depression, autism spectrum disorder, insomnia, mild cognitive impairment, etc. (Mild to moderate treated ADD/ADHD, anxiety, and/or depression are allowed.)
* Score on the Montreal Cognitive Assessment (MoCA) <23
* Score on the Generalized Anxiety Disorder-7 Scale ≥ 10
* Score on the Patient Health Questionnaire-2 ≥ 2 and score on the Patient Health Questionnaire-9 ≥ 10
* Any current (within last 3 month) or chronic medical conditions, including any musculoskeletal, cardiovascular, pulmonary, metabolic, psychiatric or neurological diagnosis that affects activities of daily living or would confound testing or place the subject at risk by participating, such as a significant cardiovascular condition or event (e.g., heart attack < 3 months ago, uncontrolled atrial fibrillation, uncontrolled angina, congestive heart failure, chronic obstructive pulmonary disorder, or peripheral vascular disease)
* Any impaired sensation or weakness in either lower extremity
* History of serious concussion or head injury, defined as a loss of consciousness for > 5 minutes and/or requiring medical treatment, or > 2 concussions over the lifespan
* Any history of acute or chronic problems with balance, any dizziness, or > 1 fall in the last 12 months
* Currently or regularly using any analgesic medications, over-the-counter remedies, or any other treatment for the purposes of pain relief (i.e., baby aspirin for heart health is allowed)
* Any current or chronic pain condition during the last year, located anywhere in the body with an intensity of > 2/10
* Allergy to capsaicin or hot peppers
* Any skin lesion, breakage or irritation in the area targeted for the painful stimulus
* Significant skin sensitivity to soaps/creams/perfumes or to heat
* Poor circulation in the area targeted for the painful stimulus
* Prior participation in a split-belt locomotor learning study in the Neuromotor Behavior Lab in the past 2 years

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Learning magnitude | End of day 1
  Step length asymmetry averaged over the last 25 strides of the practice period on day 1.
Retention magnitude | Beginning of day 2.
  Step length asymmetry averaged over the first 4 strides of the re-adaptation period on day 2.
Forgetting index | End of day 1 and beginning of day 2.
  Difference between retention magnitude and learning magnitude.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Morton, Principal Investigator — University of Delaware
Locations (1):
- Health Sciences Complex, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No